CLINICAL TRIAL: NCT02261506
Title: Bacteremia Antibiotic Length Actually Needed for Clinical Effectiveness: A Pilot RCT
Acronym: BALANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Kingston Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nick Daneman, Clinician Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 187-2014
Record Dates: First submitted 2014-09-26; First posted 2014-10-10 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Bacteremia
Keywords: Intensive care; bacteremia; bloodstream infection; antimicrobial; mortality; antimicrobial stewardship
MeSH Terms: conditions — Bacteremia; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 7 days (Active Comparator): Patients in 7 day arm will receive adequate antibiotics until the end of day 7 only
  Interventions: Other: 7 days of adequate antibiotic treatment durations
- 14 days (Active Comparator): Patients in 14 day arm will receive adequate antibiotics until the end of day 14 only
  Interventions: Other: 14 days of adequate antibiotic treatment durations

INTERVENTIONS:
Other: 7 days of adequate antibiotic treatment durations — We will not be randomizing patients to any specific antibiotic regimen. Patients will be randomized to fixed durations of adequate treatment: 7 versus 14 days. The selection of antibiotic(s) will be at the discretion of the treating team, although the research team will check to ensure that the selected antibiotics have an 'adequate' spectrum of coverage for the bacterial pathogen(s) isolated in the blood culture.
  Arms: 7 days
Other: 14 days of adequate antibiotic treatment durations
  Arms: 14 days

SUMMARY:
Bacteremia is a leading cause of mortality and morbidity in critically ill adults. Although bacteria in the bloodstream (bacteremia) may arise from variable infectious foci (most commonly central vascular catheter related, lung, urinary tract, intra-abdominal, or skin and soft tissue sources), because of the high attendant morbidity and mortality of bacteremia, these patients collectively represent a critically important group to study.

The consequences of the excessive antimicrobial use for individual patients, range from rash, gastrointestinal upset and diarrhea, to anaphylaxis, neutropenia, renal failure, toxic epidermal necrolysis, death, and a marked increase in ICU and hospital drug costs. One particularly concerning complication, Clostridium difficile infection, has increased in incidence and severity over the past decade. Much of this burden could be prevented through reduction in unnecessary antibiotic use.

Another major consequence of excessive antibiotic use is antimicrobial resistance. Antibiotic resistance is not only a concern for the patient who receives antibiotics, but also for neighbouring patients in the ICU, as well as future patients in the ICU and the hospital at large - through patient-to-patient transmission, and environmental contamination.

No previous randomized controlled trials have directly compared shorter versus longer durations of antimicrobial treatment in these patients. The investigators will conduct a multi-center randomized concealed allocation trial of shorter duration (7 days) versus longer duration (14 days) antibiotic treatment for critically ill patients with bacteremia admitted to ICU. Eligible, patients will be randomized to either 7 days or 14 days of adequate antimicrobial treatment. The selection of type, dose and route of antibiotics will be at the discretion of the treating physicians, but the duration of treatment (7 versus 14 days) will be determined by randomization group. The randomization assignment will not be communicated to the study research coordinator, study critical care or infectious diseases investigators or clinicians until day 8. The primary outcome for the main trial will be 90-day mortality.

The study will be initiated at Sunnybrook Health Sciences Centre in Toronto, Ontario, and then rolled out to a second site at Kingston General Hospital in Kingston, Ontario. These sites will be sufficient to meet the sample size goals for the pilot RCT, but if additional funds are obtained the investigators will also roll out to the other Canadian ICUs listed below. The goal of adding these additional sites will be to increase the generalizability of the findings with respect to trial feasibility

ELIGIBILITY:
Inclusion Criteria:

* Patient is in the ICU at time the blood culture result reported as positive AND
* Patient has a positive blood culture with pathogenic bacteria.

Exclusion Criteria:

* Patient already enrolled in the trial
* Patient has severe immune system compromise, as defined by: absolute neutrophil count <0.5x109/L; or is receiving immunosuppressive treatment for solid organ or bone marrow or stem cell transplant
* Patient has syndrome with well-defined requirement for prolonged treatment:

  * infective endocarditis
  * osteomyelitis/septic arthritis
  * undrainable/undrained abscess
  * unremovable/unremoved prosthetic-associated infection
* Patient has a single positive blood culture with a common contaminant organism according to Clinical Laboratory & Standards Institute (CLSI) Guidelines: coagulase negative staphylococci; or Bacillus spp.; or Corynebacterium spp.; or Propionobacterium spp.; or Aerococcus spp.; or Micrococcus spp.
* Patient has a positive blood culture with Staphylococcus aureus.
* Patient has a positive blood culture with Candida spp. or other fungal species.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Adherence to treatment duration protocol (proportion of treatment courses) | 15 days
  We will consider the main trial to be feasible and worthy of embarking on a larger mortality-powered RCT if 90% of antibiotic treatment courses are within 7± 2 days in the shorter duration treatment arm or 14 ± 2 days in the longer duration treatment arm.
Rate of recruitment (patients per site, per month) | For up to 1 year
  We will consider the main trial to be feasible if we achieve recruitment rates of at least 1 patient per 4 weeks, on average, per participating site.

SECONDARY OUTCOMES:
ICU mortality | Recorded as alive or dead at ICU discharge following index positive blood culture for an expected average of 2 weeks assesses upto one year.
Hospital mortality | recorded as alive or dead at hospital discharge following index positive blood culture for an expected average of 4 weeks assesses upto one year.
90 day mortality | Recorded as alive or dead at 90 days following index positive blood culture
Relapse rates of bacteremia | Upto 30 days after adequate antibiotic treatment
  Defined as the recurrence of bacteremia due to original infecting organism (same Genus and species) after documentation of negative blood cultures or clinical improvement and within 30 days after completing course of adequate antimicrobial therapy.
Antibiotic allergy | Up to 30 days from start of antibiotic treatment.
  Effect of medication on body that produces the allergic reaction to a medication like:
  * Hives
  * Itching of the skin or eyes
  * Skin rash
  * Swelling of the lips, tongue, or face
  * Wheezing
Anaphylaxis | Up to 30 days from start of antibiotic treatment
  To be considered anaphylaxis, the patient must have had >=1 of the following 3 criteria that a medical team member attributed to an Antimicrobial
  * Acute onset of skin or mucosal tissue changes (hives, itching/flush, lip/tongue/uvula swelling) over minutes/hours, accompanied by
    * respiratory compromise (dyspnea, wheeze, stridor, hypoxemia), AND/OR
    * reduced blood pressure or symptoms/signs of end organ dysfunction from shock
  * Rapid onset of two or more of the following
    * involvement of the skin-mucosa (hives, itch//flush, swollen lips/tongue/uvula)
    * respiratory compromise
    * reduced BP or associated symptoms/signs
    * persistent gastrointestinal symptoms/signs (crampy abdominal pain, vomiting)
  * Reduced blood pressure after exposure to a known allergen for that patient
Antimicrobial-related acute kidney injury | Up to 30 days from start of antibiotic treatment
  To be considered Antimicrobial-associated renal injury, a medical team member must have attributed the renal injury to the Antimicrobial, and the severity of the renal injury must meet one of these (RIFLE criteria):
  * Risk: GFR decrease >25%, serum creatinine increased 1.5 times or urine production of <0.5 ml/kg/hr for 6 hours
  * Injury: GFR decrease >50%, doubling of creatinine or urine production <0.5 ml/kg/hr for 12 hours
  * Failure: GFR decrease >75%, tripling of creatinine or creatinine >355 μmol/l (with a rise of >44) (>4 mg/dl) OR urine output below 0.3 ml/kg/hr for 24 hours
  * Loss: persistent AKI or complete loss of kidney function for more than 4 weeks
  * End-stage renal disease: need for renal replacement therapy (RRT) for more than 3 months
Antimicrobial-related hepatitis | Up to 30 days from start of antibiotic treatment
  To be considered Antimicrobial-associated hepatitis, a medical team member must have attributed the hepatitis to the Antimicrobial, and the severity of the hepatitis must meet this FDA criteria for hepatic adverse events:
  o ALT> 3x the upper limit of normal
Rates of Clostridium difficile infection in hospital | Upto 30 days after index blood culture collection date
  Defined as a positive PCR or ELISA test for Clostridium difficile toxin in the context of diarrhea within hospital of bacteremia diagnosis.
Rates of secondary nosocomial infection with antimicrobial resistant organisms in hospital | Upto 30 days after index blood culture collection date
ICU lengths of stay | For the duration of ICU stay, expected for an average of 30 days assessed up to 1 year.
Hospital lengths of stay | For the duration of Hospital stay, expected for an average of 30 days assessed up to 1 year.
Mechanical ventilation duration | For the duration of ICU and Hospital stay, expected for an average of 30 days
  Defined as the number of consecutive days receiving invasive (via an endotracheal tube or tracheostomy), or non-invasive (via a facemask, nasal mask, or helmet) ventilation. Durations will be calculated for all patients then separately for patients who died within hospital and those who did not die.
Vasopressor duration in ICU | For the duration of ICU and Hospital stay, expected for an average of 30 days
  Defined as the number of consecutive days receiving intravenous vasoactive medications (e.g. epinephrine, norepinephrine, vasopressin, dopamine, phenylephrine, dobutamine, milrinone). Durations will be calculated for all patients then separately for patients who died within hospital and those who did not die.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Daneman, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (17):
- Canada (17):
  - Foothills Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II Hospital, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - CHUM, Montreal, Quebec
  - Centre hospitalier affilié universitaire de Québec, Québec, Quebec
  - CSSS de Trois-Rivières, Québec, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Derived] Daneman N, Rishu AH, Pinto R, Aslanian P, Bagshaw SM, Carignan A, Charbonney E, Coburn B, Cook DJ, Detsky ME, Dodek P, Hall R, Kumar A, Lamontagne F, Lauzier F, Marshall JC, Martin CM, McIntyre L, Muscedere J, Reynolds S, Sligl W, Stelfox HT, Wilcox ME, Fowler RA; Canadian Critical Care Trials Group. 7 versus 14 days of antibiotic treatment for critically ill patients with bloodstream infection: a pilot randomized clinical trial. Trials. 2018 Feb 17;19(1):111. doi: 10.1186/s13063-018-2474-1. PMID 29452598
- [Derived] Daneman N, Rishu AH, Xiong W, Bagshaw SM, Cook DJ, Dodek P, Hall R, Kumar A, Lamontagne F, Lauzier F, Marshall JC, Martin CM, McIntyre L, Muscedere J, Reynolds S, Stelfox HT, Fowler RA; Canadian Critical Care Trials Group. Bacteremia Antibiotic Length Actually Needed for Clinical Effectiveness (BALANCE): study protocol for a pilot randomized controlled trial. Trials. 2015 Apr 18;16:173. doi: 10.1186/s13063-015-0688-z. PMID 25903783